CLINICAL TRIAL: NCT06557174
Title: A Phase Ib/III Multi-center, Randomized and Positive Control Study to Evaluate IMC-002 Safety and Efficacy in in Neuromyelitis Optica Spectrum Disorder (NMOSD) Patients
Brief Title: A Study to Evaluate IMC-002 in Neuromyelitis Optica Spectrum Disorder (NMOSD) Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmuneCare Biopharmaceuticals (Shanghai) Co., Ltd. (Other)
Responsible Party: Sponsor
Organization: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMC002-N-01
Record Dates: First submitted 2024-08-11; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Neuromyelitis Optica Spectrum Disorder (NMOSD)
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMC-002 (Experimental): intravenous injection of 0.8mg/kg、1.2mg/kg
  Interventions: Drug: IMC-002
- mycophenolate mofetil， MMF (Active Comparator): mycophenolate mofetil will be administrated as monotherapy control for 0.2g daily oral.
  Interventions: Drug: mycophenolate mofetil， MMF

INTERVENTIONS:
Drug: IMC-002 — intravenous injection: Weekly administered for a period of first 4 weeks, then rest for 20 weeks. After the administration of the testing drug, if the subject's symptoms get worsen, a rescue therapy need to be adopted as based on Investigator's judgement, the testing drug injection should be discontinued.
  Arms: IMC-002
Drug: mycophenolate mofetil， MMF — daily oral 0.2g
  Arms: mycophenolate mofetil， MMF

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of IMC-002 in the treatment of NMOSD.

DETAILED DESCRIPTION:
This is a phase Ib/III study, including 2 stage, phase Ib study to find the dose for phase II study between 0.8mg/kg、1.2mg/kg dose level, Phase III study is a multi-center, randomized, double-blind, positive control study to evaluate the safety and efficacy of IMC-002 in Neuromyelitis Optica Spectrum Disorder (NMOSD)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years, inclusive, at the time of informed consent
* Have a diagnosis of AQP4 antibody seropositive NMOSD according to the International Panel for NMO Diagnosis (IPND) criteria
* Confirmation of NMOSD diagnosis with AQP4+ antibodies
* The EDSS score should be ≤7.0
* Have clinical evidence of at least 1 documented attack or relapse (including first attack) in the last 2 years prior to screening

Exclusion Criteria:

* Have received rituximab or other anti-CD20 drugs treatment within 6 months
* Have been used any monoclonal antibodies or research drugs for immunomodulatory effects within 3 months or within 5 half-life periods of the drug.
* Females who are pregnant or lactating.
* Have active infection at screening, or recent serious infection (i.e., requiring intravenous antimicrobial therapy or hospitalization) ; history of or existing infection of human immunodeficiency virus(HIV), hepatitis C virus (HCV), or Mycobacterium tuberculosis. Patients must have negative test results for HCV antibody, HIV 1 and HIV 2 antibodies, and a mycobacterium tuberculosis test (test method to be determined).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of relapse-free patients | Up to Week 24

SECONDARY OUTCOMES:
Time to first relapse (TFR) | Up to Week 24
Mean change from baseline in Expanded Disability Status Scale (EDSS) score over the course of the study | Baseline (Day -28 to Day -1) to Week 24
  The Expanded Disability Status Scale ranges from 0 to 10 in 0.5 unit increments. Higher results represent higher levels of disability